CLINICAL TRIAL: NCT04325711
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of CSPCHA131 in Patients With Advanced Solid Tumors
Brief Title: A Study of CSPCHA131 in Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPCHA131-CSP-001
Record Dates: First submitted 2020-03-10; First posted 2020-03-30 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CSPCH131 dose Escalation and expansion (Experimental): In the dose escalation part of Stage I, five dose levels will be tested according to the "3 + 3" dose-escalation design. Whether and how to carry out the follow-up study parts will be decided by the PI and sponsor on the basis of the achieved results of safety, tolerability and effectiveness of CSPCHA131.
  Interventions: Drug: CSPCHA131

INTERVENTIONS:
Drug: CSPCHA131 — CSPCHA131 will be administered twice weekly in the first three weeks of a 4-week cycle.

SUMMARY:
The study was designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of CSPCHA131 alone or plus chemotherapy in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a dose escalation and expansion study with the aim to evaluate and characterize the tolerability and safety profile of CSPCHA131 alone (Stage I) or plus chemotherapy (Stage II) in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1.18-75 years of age.
* 2. Histologically or cytologically confirmed diagnosis of advanced or metastatic malignant solid tumors, for which standard therapy either does not exist or has been proven ineffective or intolerable for the patient.
* 3. At least one measurable tumor lesion according to RECIST version 1.1.
* 4. ECOG performance status of 0 or 1.
* 5. Life expectancy ≥ 3 months. No cardiac insufficiency or serious abnormalities in the electrocardiogram at baseline.

Exclusion Criteria:

* 1. Administration of chemotherapy, radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy, other anti-tumor treatments or an investigational drug within 4 weeks or 5 half-lives, whichever is longer, preceding the first dose of study treatment.
* 2. Have undergone surgery within 4 weeks prior to the study treatment or have not fully recovered from any previous invasive procedure.
* 3. Adverse reactions to previous anti-tumor treatments that levels have not recovered to grade 1 or less.
* 4. Patients with evidence of uncontrolled nervous system metastasis or meningeal metastases, in the opinion of the investigator, not suitable for enrollment.
* 5. Active infections of grade 2 or above.
* 6. Peripheral neuropathy of grade 2 or above.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-04-12 (Estimated); Study Completion 2021-04-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and incidence of dose limiting toxicity (DLT) within the first cycle at each dose level. | Time Frame: 28 days
Incidence of adverse events (AEs) and serious adverse events throughout the trial; | from enrollment to the end of the trial (2 years)

SECONDARY OUTCOMES:
Objective response rate (ORR) defined by RECIST Criteria Version 1.1; | from enrollment to the end of the trial (2 years)
  ORR is defined as the proportion of patients who achieve complete response (CR) or partial response (PR).
Progression free survival (PFS) defined by RECIST Criteria Version 1.1; | from enrollment to the end of the trial (2 years)
  PFS is defined as the time from the start of treatment until disease progression or death from any cause, whichever is earlier.
AUC0-t | 28 days
  PK parameter: AUC0-t
AUC0-∞ | 28 days
  PK parameter: AUC0-∞
Cmax | 28 days
  PK parameter: Cmax
Css_max | 28 days
  PK parameter: Css_max
Css_min | 28 days
  PK parameter: Css_min
DF | 28 days
  PK parameter: DF
Ke | 28 days
  PK parameter: Ke
Tmax | 28 days
  PK parameter: Tmax
Vz | 28 days
  PK parameter: Vz
T1/2 | 28 days
  PK parameter: T1/2
CL | 28 days
  PK parameter: CL

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China